CLINICAL TRIAL: NCT06463496
Title: Balance and Executive Function in Middle-age and Older Patients With Heart Failure in Post-Acute Care Program
Status: Active, not recruiting | Type: Observational
Sponsor: Chang Chia-Jung (Other)
Collaborators: Kaohsiung Veterans General Hospital. (Other)
Responsible Party: Sponsor-Investigator, Chang Chia-Jung, Occupational therqapy, Kaohsiung Veterans General Hospital.
Organization: Kaohsiung Veterans General Hospital. (Other)
Other Study IDs: KSVGH24-CT6-08
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Heart Failure
Keywords: Heart Failure; Balance Function; Executive Function
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Heart failure group: Patients with heart failure in post-acute care program
- Healthy control group: The age- and gender-matched healthy control group

SUMMARY:
This trial is a single-center clinical trial in Taiwan with an expected enrollment of 60 people in Taiwan. The purpose of this trial is to compare the performance of middle-aged and elderly patients with subacute heart failure with that of a healthy control group in terms of balance function and executive function, as well as to investigate whether there is a correlation between balance function and executive function in middle-aged and elderly patients with heart failure and to track the changes in balance and executive function one month and three months after discharge from the hospital. Please think carefully before deciding whether to participate in this trial.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with heart failure and receiving post-acute care program for heart failure
* Left ventricular ejection fraction≦40%
* Age ≥ 45
* No cognitive impairment
* Ambulate independently or with the use of aids
* Clinical symptoms are stable
* Voluntary participation

Exclusion Criteria:

* Use of medications that cause dizziness or interfere with balance
* Have other diagnoses that may affect balance, such as stroke, Parkinson's disease
* Color blindness, severe hearing or visual impairment that prevents reading questions and listening to instructions

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 1. Middle-aged and older patients with heart failure in in Post-Acute Care Program
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-06-17 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-02-28 (Estimated)

PRIMARY OUTCOMES:
Berg Balance Scale | T0 : Baseline ； T1: one month after discharge； T2: three months discharge
  The balance function will be evaluated using the Berg Balance Scale. Berg Balance Scale have 14 subtests, each of which is scored on a scale of 0 to 4, for a total score of 56, with higher scores indicating better balance.
Timed Up and Go Test | T0 : Baseline ； T1: one month after discharge； T2: three months discharge
  The balance function will be evaluated using the Timed Up and Go Test. Timed Up and Go Test use a chronograph to measure the total time spent (in seconds), with less time representing better ability.

SECONDARY OUTCOMES:
Color Trails Test | T0 : Baseline ； T1: one month after discharge； T2: three months discharge
  The Working memory will be evaluated using Color Trails Test. Scoring is based on the total number of seconds to complete the test. Lower scores represent greater difficulty inWorking memory .
The Stroop Color and Word Test | T0 : Baseline ； T1: one month after discharge； T2: three months discharge
  The Inhibitor Control will be evaluated using the Stroop Color and Word Test. The test consisted of three parts, each spanning 45 s where participants read out as many colour words such as ''red, green, blue and purple'' or coloured items words as possible.
  Number of items corrected and wrongly read out were used to compute the predicted colour-word (Pcw) and interference (IF).Lower scores represent greater difficulty in inhibiting incongruence.
Digit Span Test | T0 : Baseline ； T1: one month after discharge； T2: three months discharge
  The Cognitive flexibility will be evaluated using the Digit Span test. The scores range from 0 to 45. Lower scores represent greater difficulty in Cognitive flexibility .

CONTACTS AND LOCATIONS:
Locations (1):
- Kaohsiung Veterans General Hospital, Kaohsiung City, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided